CLINICAL TRIAL: NCT05662722
Title: Use of Infrared Thermography in the Measurement of Facial Blood Flow After the Application of Percutaneous Needle Electrolysis (PNE) on the Concha of the Ear
Brief Title: Percutaneous Needle Electrolysis (PNE) on the Concha of the Ear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEID/2022/2/028
Record Dates: First submitted 2022-12-06; First posted 2022-12-22 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: clinical random assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple (care provider, evaluator and outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pecutaneous electrolysis group (Experimental): Subjects were treated twice (one day and one week). The technique consisted in the application of a galvanic electrical current using a needle as an electrode that will be inserted into the concha of the ear. The subjects were lying in supinus.
  Interventions: Other: percutaneous needle electrolysis
- dry needling group (Other): Subjects were treated twice (one day and one week). The technique consisted in the puncture with a needle in the concha of the ear. The subjects were lying in supinus.
  Interventions: Other: Dry needling
- Sham group (Sham Comparator): Subjects were treated twice (one day and one week). The technique consisted in the puncture with a sham-needle in the concha of the ear. The subjects were lying in supinus.
  Interventions: Other: Sham needling

INTERVENTIONS:
Other: percutaneous needle electrolysis — It´s an intervention of physiotherapy. It´s an invasive technique.
  Arms: Pecutaneous electrolysis group
Other: Dry needling — It´s an intervention of physiotherapy. It´s an invasive technique.
  Arms: dry needling group
Other: Sham needling — It´s an intervention of physiotherapy. It´s an invasive technique simulation.
  Arms: Sham group

SUMMARY:
Headache is a very frequent symptom among the world population, the adult population with an active headache disorder are 46% for headache in general, 11% for migraine, 42% for tension-type headache and 3% for chronic daily headache. There are different therapeutic approaches for the improvement of headache. Transcutaneous stimulation of the auricular vagal nerve is being used for the treatment of headache due to the involvement of the vagus nerve in inflammation and pain modulation. On the other hand, galvanic current has shown a measurable effect by increasing parasympathetic activity. The objective of this clinical trial is to stimulate the auricular vagal nerve with galvanic current using a needle as an electrode that will be inserted into the concha of the ear. As a tool for measuring results, infrared thermography will be used to observe changes in facial skin temperature, since patients with high sympathetic activity present a characteristic pattern of "cold nose" and/or "cold patch". In addition, variables that record changes in autonomic activity such as skin conductance and heart rate variability will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Headache with a frequency of at least one monthly episode.
* Present the "cold nose" and/or "cold patch" pattern

Exclusion Criteria:

* Do not present a "cold nose" and/or "cold patch" pattern
* Pregnant women
* Subjects with facial alterations that may affect facial vascularization (sinusitis, allergies...)
* Patients with belonephobia or allergy to metals or any material used in the procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Skin temperature | Change from Baseline up to 30 minutes
  It´s a camera to take infrared thermal images. The images provide facial temperature measurement.
Headache Impact Test (HIT-6) | Change from Baseline up to 30 minutes
  Headache Impact (HIT) is a tool used to measure the impact headaches have on your ability to function at work, home, school and in social situations. Your score shows you the effect that headaches they have in normal daily life and in their ability to function.A score of 60 or higher is associated with a very severe impact. A score equal to or less than 49 is associated with a low impact.

SECONDARY OUTCOMES:
Skin bioimpedance | Change from Baseline up to 30 minutes
  It´s a system to acquire bio-electrical and physiological signals (galvanic skin conductance, heart rate variability), and transfer these signals to a computer for processing an analysis.
Heart rate variability | Change from Baseline up to 30 minutes
  It´s a system to acquire bio-electrical and physiological signals (galvanic skin conductance, heart rate variability), and transfer these signals to a computer for processing an analysis.
Numerical Rating Scale | Change from Baseline up to three months
  Patients vebally requested to rate their pain: "Rate your pain from = (no pain) to 10 (unbearable pain)
Patients global impressions scale: | Change from Baseline up to three months
  It´s the Patient reported outcomes counterpart to the Clinical Global Impressions scale. The PGIS are 1-item questionnaire that ask an individual patient to rate the severity of a specific condition (single-state scales) at baseline and or to rate at endpoint the perceived change in is/her condition in response to therapy; in the other hand PGIC measures change in clinical status.
Pittsburg Sleep Quality Index score | Change from Baseline up to three months
  Improvement in Pittsburg Sleep Quality Index (PSQI), Scale is 0 to 21, higher score is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Principal Investigator — Alcala University
Locations (1):
- Physioterapy and Pain center research, Alcalá de Henares, Madrid, Spain